CLINICAL TRIAL: NCT02909920
Title: Effectiveness of Telerehabilitation Program Following Surgery Procedures in Subacromial Syndrome Compared With Traditional Therapy. A Randomized Clinical Trial (Telerehab)
Brief Title: Effectiveness of Telerehabilitation Program in Subacromial Syndrome (Telerehab Sis)
Acronym: telerehab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jose Manuel Pastora Bernal (Other)
Collaborators: University of Malaga (Other); Hospital Costa del Sol (Other)
Responsible Party: Sponsor-Investigator, Jose Manuel Pastora Bernal, MSc Research in Health Sciences (Phd Health Sciences Student), University of Malaga
Organization: University of Malaga (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0761-M1-16
Record Dates: First submitted 2016-09-14; First posted 2016-09-21 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Telerehabilitation; Physiotherapy; Surgery; Telemedicine
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telerehabilitation (Experimental): The Telerehabilitation group receives a standardized and customized exercises through a web application that allows the Physiotherapist generate videos, images and parameters of each exercise program and send them via email for each patient. Patients are initially supervised by a physiotherapist who will conduct videoconference sessions to ensure proper execution of exercises and encourage patient adherence.
  Interventions: Other: Telerehabilitation
- Traditional Physiotherapy (Active Comparator): Traditional Physiotherapy group receives assistance in a physiotherapy center through the usual procedure of rehabilitation in Spain consisting in personalized therapy 1 to 1 with a physical therapist and exercise programs for home.
  Interventions: Other: Traditional Physiotherapy

INTERVENTIONS:
Other: Telerehabilitation — Initial Videoconference following telerehabilitation programs self-workout exercise with video support.
  Arms: Telerehabilitation
Other: Traditional Physiotherapy — Traditional Physiotherapy receives assistance in a physiotherapy center with personalized therapy consisting of 1 to 1 with a physical therapist (Manual Therapy, home exercise programs and other physiotherapy techniques).
  Arms: Traditional Physiotherapy

SUMMARY:
Shoulder pain is a common and high prevalence in the general population. Subacromial Syndrome (Shoulder Impingement Syndrome (SIS)) is the most frequent cause. SIS patients suffering pain, muscle weakness and loss of movement in the affected joint. Initial treatment of the SIS is predominantly conservative. Surgical option has high success rates and is often used when conservative strategy fails. Traditional Physiotherapy and Postoperative exercises is needed to the recovery of joint range, muscle strength, stability and functionality. This Research evaluates the feasibility and effectiveness of a telerehabilitatión Program in SIS after surgery compared with traditional therapy.

DETAILED DESCRIPTION:
In addition to traditional physiotherapy, Telerehabilitation programs have proven their effectiveness, validity, noninferiority and important advantages in various neurological, cognitive diseases and musculoskeletal disorders; meaning an opportunity to define new social and intervention policies.

Subjects are randomly assigned to 1) Telerehabilitation Group 2) Traditional Therapy Group. After randomization, patients in both groups received an initial evaluation. Data will be collected by a blinded evaluator.

The Telerehabilitation group receives a standardized and customized exercises to perform, through a web application that allows the Physiotherapist generate videos, images and parameters of each exercise program and send them via email for each patient.

Telerehabilitation program describes the exercises to be performed, the number of repetitions depending on the level of training and criteria for progression.

Patients are initially supervised by a physiotherapist who will conduct three training sessions through individual videoconference, to ensure proper execution of exercises and encourage patient adherence. Patients are instructed to perform self-workout video exercises following Telerehabilitation program as well as a supporting document we call Telerehabilitation Manual Patient.

Traditional group receives assistance in a physiotherapy center through the usual procedure of rehabilitation in Spain, personalized therapy consisting of 1 to 1 with a physical therapist and exercise programs at home.

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18 and 65 years
* Subacromial Syndrome Diagnosis ICD-9 CM 726.10, 726.12, 726.19 issued by specialist in Orthopaedic Surgery and Rehabilitation Specialist
* Receive Surgical Procedure (arthroscopy or open approach (subacromial decompression with partial acromioplasty, with or without coracoacromial release) and prescription of rehabilitation process.
* He lives in Spain during the investigation period
* Provides in home computer with internet technology (personal computer, laptop, tablet or Smartphone)
* Skills and knowledge to access email

Exclusion Criteria:

* Previously Surgery intervention in same shoulder.
* Patients receiving non-surgical procedure based on the recommendations for Subacromial Syndrome
* Unfit cognitive ability to use technological tools

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Changes in Simple Shoulder Test (SST) score | Initial, 4 weeks, 8 weeks and 12 weeks
  Simple Shoulder Test is a validated instrument that features 12 one-dimensional answers questions with dichotomous (Yes / No). It is a short questionnaire (2-3 minutes), easy to understand and fulfill what gives validity and comparability with other subjective questionnaires. The total score of 12 questions (2 related to pain, 7 on the force, and 3 on the range of motion) where 0 is the worst result and 100 if the best shoulder function is measured, calculated based on the number of positive responses multiplied by 100. questionnaire. The internal consistency of the test was measured by Cronbach's alpha = 0.85. We will assess changes in this test score.

SECONDARY OUTCOMES:
Changes in Constant Shoulder test Score | Initial, 4 weeks, 8 weeks and 12 weeks
  Constant score is an assessment tool universally used and accepted for shoulder function. It includes a subjective assessment of pain and ability to perform daily activities (work, sport, dream and positioning of the hand in space), and an objective assessment of mobility and strength through physical examination. We will assess changes in this test score.

OTHER OUTCOMES:
Telemedicine Satisfaction and Usefulness Questionnaire (TSUQ) (Spanish adaptation) | 12 weeks
  Acceptance and usability of telemedicine applications is a prerequisite for identifying potential clinical benefits of this technology. Consequently, it is important to supplement this research with tools to examine the satisfaction and perception of patients.
Direct and Indirect Costs | 12 weeks
  This economic analysis is based on the perspective of the health sector, which means that only those for health interventions costs will be considered, and unrelated costs for the patient. Therefore, only the costs associated with the provision of health services in the traditional physiotherapy group telerehabilitación be taken into account.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Manuel Pastora Bernal, Principal Investigator — University of Malaga; Rocio Martín Valero, Study Director — University of Malaga; Francisco Javier Barón López, Study Director — University of Malaga
Locations (1):
- Faculty of Health Sciences Universidad de Málaga, Málaga, Malaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luime JJ, Koes BW, Hendriksen IJ, Burdorf A, Verhagen AP, Miedema HS, Verhaar JA. Prevalence and incidence of shoulder pain in the general population; a systematic review. Scand J Rheumatol. 2004;33(2):73-81. doi: 10.1080/03009740310004667. PMID 15163107
- [Background] Michener LA, Walsworth MK, Burnet EN. Effectiveness of rehabilitation for patients with subacromial impingement syndrome: a systematic review. J Hand Ther. 2004 Apr-Jun;17(2):152-64. doi: 10.1197/j.jht.2004.02.004. PMID 15162102
- [Background] Ludewig PM, Cook TM. Alterations in shoulder kinematics and associated muscle activity in people with symptoms of shoulder impingement. Phys Ther. 2000 Mar;80(3):276-91. PMID 10696154
- [Background] Senbursa G, Baltaci G, Atay A. Comparison of conservative treatment with and without manual physical therapy for patients with shoulder impingement syndrome: a prospective, randomized clinical trial. Knee Surg Sports Traumatol Arthrosc. 2007 Jul;15(7):915-21. doi: 10.1007/s00167-007-0288-x. Epub 2007 Feb 28. PMID 17333123
- [Background] Marin-Gomez M, Navarro-Collado MJ, Peiro S, Trenor-Gomis C, Paya-Rubio A, Bernal-Delgado E, Hernandez-Royo A. [The quality of care in shoulder pain. A medical audit]. Gac Sanit. 2006 Mar-Apr;20(2):116-23. doi: 10.1157/13087322. Spanish. PMID 16753088
- [Background] Virta L, Joranger P, Brox JI, Eriksson R. Costs of shoulder pain and resource use in primary health care: a cost-of-illness study in Sweden. BMC Musculoskelet Disord. 2012 Feb 10;13:17. doi: 10.1186/1471-2474-13-17. PMID 22325050
- [Background] Matsen FA AC. Subacromial impingement. In: Rockwood CA, Matsen FA, eds. Shoulder Philadelphia, Pa WB Saunders Co; 1990623-646.
- [Background] van der Windt DA, Koes BW, de Jong BA, Bouter LM. Shoulder disorders in general practice: incidence, patient characteristics, and management. Ann Rheum Dis. 1995 Dec;54(12):959-64. doi: 10.1136/ard.54.12.959. PMID 8546527
- [Background] Meister K. Internal impingement in the shoulder of the overhand athlete: pathophysiology, diagnosis, and treatment. Am J Orthop (Belle Mead NJ). 2000 Jun;29(6):433-8. PMID 10890456
- [Background] Walther M, Werner A, Stahlschmidt T, Woelfel R, Gohlke F. The subacromial impingement syndrome of the shoulder treated by conventional physiotherapy, self-training, and a shoulder brace: results of a prospective, randomized study. J Shoulder Elbow Surg. 2004 Jul-Aug;13(4):417-23. doi: 10.1016/j.jse.2004.02.002. PMID 15220882
- [Background] Fongemie AE, Buss DD, Rolnick SJ. Management of shoulder impingement syndrome and rotator cuff tears. Am Fam Physician. 1998 Feb 15;57(4):667-74, 680-2. PMID 9490991
- [Background] Michener LA, McClure PW, Karduna AR. Anatomical and biomechanical mechanisms of subacromial impingement syndrome. Clin Biomech (Bristol). 2003 Jun;18(5):369-79. doi: 10.1016/s0268-0033(03)00047-0. PMID 12763431
- [Background] Hegedus EJ, Goode A, Campbell S, Morin A, Tamaddoni M, Moorman CT 3rd, Cook C. Physical examination tests of the shoulder: a systematic review with meta-analysis of individual tests. Br J Sports Med. 2008 Feb;42(2):80-92; discussion 92. doi: 10.1136/bjsm.2007.038406. Epub 2007 Aug 24. PMID 17720798
- [Background] Chaudhury S, Gwilym SE, Moser J, Carr AJ. Surgical options for patients with shoulder pain. Nat Rev Rheumatol. 2010 Apr;6(4):217-26. doi: 10.1038/nrrheum.2010.25. PMID 20357791
- [Background] Gebremariam L, Hay EM, Koes BW, Huisstede BM. Effectiveness of surgical and postsurgical interventions for the subacromial impingement syndrome: a systematic review. Arch Phys Med Rehabil. 2011 Nov;92(11):1900-13. doi: 10.1016/j.apmr.2011.06.006. PMID 22032225
- [Background] Checroun AJ, Dennis MG, Zuckerman JD. Open versus arthroscopic decompression for subacromial impingement. A comprehensive review of the literature from the last 25 years. Bull Hosp Jt Dis. 1998;57(3):145-51. PMID 9809180
- [Background] Klintberg IH, Svantesson U, Karlsson J. Long-term patient satisfaction and functional outcome 8-11 years after subacromial decompression. Knee Surg Sports Traumatol Arthrosc. 2010 Mar;18(3):394-403. doi: 10.1007/s00167-009-0963-1. Epub 2009 Oct 23. PMID 19851753
- [Background] Coghlan JA, Buchbinder R, Green S, Johnston RV, Bell SN. Surgery for rotator cuff disease. Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD005619. doi: 10.1002/14651858.CD005619.pub2. PMID 18254085
- [Background] Hultenheim Klintberg I, Gunnarsson AC, Styf J, Karlsson J. Early activation or a more protective regime after arthroscopic subacromial decompression--a description of clinical changes with two different physiotherapy treatment protocols--a prospective, randomized pilot study with a two-year follow-up. Clin Rehabil. 2008 Oct-Nov;22(10-11):951-65. doi: 10.1177/0269215508090771. PMID 18955427
- [Background] Christiansen DH, Frost P, Falla D, Haahr JP, Frich LH, Andrea LC, Svendsen SW. Effectiveness of Standardized Physical Therapy Exercises for Patients With Difficulty Returning to Usual Activities After Decompression Surgery for Subacromial Impingement Syndrome: Randomized Controlled Trial. Phys Ther. 2016 Jun;96(6):787-96. doi: 10.2522/ptj.20150652. Epub 2016 Feb 25. PMID 26916927
- [Background] Russell TG. Physical rehabilitation using telemedicine. J Telemed Telecare. 2007;13(5):217-20. doi: 10.1258/135763307781458886. PMID 17697506
- [Background] Lathan CE, Kinsella A, Rosen MJ, Winters J, Trepagnier C. Aspects of human factors engineering in home telemedicine and telerehabilitation systems. Telemed J. 1999 Summer;5(2):169-75. doi: 10.1089/107830299312131. PMID 10908429
- [Background] Winters JM. Telerehabilitation research: emerging opportunities. Annu Rev Biomed Eng. 2002;4:287-320. doi: 10.1146/annurev.bioeng.4.112801.121923. Epub 2002 Mar 22. PMID 12117760
- [Background] Marshall SG, Shaw DK, Honles GL, Sparks KE. Interdisciplinary approach to the rehabilitation of an 18-year-old patient with bronchopulmonary dysplasia, using telerehabilitation technology. Respir Care. 2008 Mar;53(3):346-50. PMID 18291051
- [Background] Seelman KD, Hartman LM. Telerehabilitation: policy issues and research tools. Int J Telerehabil. 2009 Sep 4;1(1):47-58. doi: 10.5195/ijt.2009.6013. eCollection 2009 Fall. PMID 25945162
- [Background] Rosen MJ. Telerehabilitation. Telemed J E Health. 2004 Summer;10(2):115-7. doi: 10.1089/tmj.2004.10.115. No abstract available. PMID 15319039
- [Background] Theodoros D, Russell T. Telerehabilitation: current perspectives. Stud Health Technol Inform. 2008;131:191-209. PMID 18431862
- [Background] Gagnon MP, Duplantie J, Fortin JP, Landry R. Implementing telehealth to support medical practice in rural/remote regions: what are the conditions for success? Implement Sci. 2006 Aug 24;1:18. doi: 10.1186/1748-5908-1-18. PMID 16930484
- [Background] Jelcic N, Agostini M, Meneghello F, Busse C, Parise S, Galano A, Tonin P, Dam M, Cagnin A. Feasibility and efficacy of cognitive telerehabilitation in early Alzheimer's disease: a pilot study. Clin Interv Aging. 2014 Sep 24;9:1605-11. doi: 10.2147/CIA.S68145. eCollection 2014. PMID 25284993
- [Background] Houlihan BV, Jette A, Friedman RH, Paasche-Orlow M, Ni P, Wierbicky J, Williams K, Ducharme S, Zazula J, Cuevas P, Rosenblum D, Williams S. A pilot study of a telehealth intervention for persons with spinal cord dysfunction. Spinal Cord. 2013 Sep;51(9):715-20. doi: 10.1038/sc.2013.45. Epub 2013 Jun 11. PMID 23752260
- [Background] Paul L, Coulter EH, Miller L, McFadyen A, Dorfman J, Mattison PG. Web-based physiotherapy for people moderately affected with Multiple Sclerosis; quantitative and qualitative data from a randomized, controlled pilot study. Clin Rehabil. 2014 Sep;28(9):924-35. doi: 10.1177/0269215514527995. Epub 2014 Apr 1. PMID 24691218
- [Background] Hoffmann T, Russell T, Thompson L, Vincent A, Nelson M. Using the Internet to assess activities of daily living and hand function in people with Parkinson's disease. NeuroRehabilitation. 2008;23(3):253-61. PMID 18560142
- [Background] Lin KH, Chen CH, Chen YY, Huang WT, Lai JS, Yu SM, Chang YJ. Bidirectional and multi-user telerehabilitation system: clinical effect on balance, functional activity, and satisfaction in patients with chronic stroke living in long-term care facilities. Sensors (Basel). 2014 Jul 11;14(7):12451-66. doi: 10.3390/s140712451. PMID 25019632
- [Background] Langan J, Delave K, Phillips L, Pangilinan P, Brown SH. Home-based telerehabilitation shows improved upper limb function in adults with chronic stroke: a pilot study. J Rehabil Med. 2013 Feb;45(2):217-20. doi: 10.2340/16501977-1115. PMID 23319181
- [Background] Deng H, Durfee WK, Nuckley DJ, Rheude BS, Severson AE, Skluzacek KM, Spindler KK, Davey CS, Carey JR. Complex versus simple ankle movement training in stroke using telerehabilitation: a randomized controlled trial. Phys Ther. 2012 Feb;92(2):197-209. doi: 10.2522/ptj.20110018. Epub 2011 Nov 17. PMID 22095209
- [Background] Jackson JC, Ely EW, Morey MC, Anderson VM, Denne LB, Clune J, Siebert CS, Archer KR, Torres R, Janz D, Schiro E, Jones J, Shintani AK, Levine B, Pun BT, Thompson J, Brummel NE, Hoenig H. Cognitive and physical rehabilitation of intensive care unit survivors: results of the RETURN randomized controlled pilot investigation. Crit Care Med. 2012 Apr;40(4):1088-97. doi: 10.1097/CCM.0b013e3182373115. PMID 22080631
- [Background] Galiano-Castillo N, Ariza-Garcia A, Cantarero-Villanueva I, Fernandez-Lao C, Diaz-Rodriguez L, Legeren-Alvarez M, Sanchez-Salado C, Del-Moral-Avila R, Arroyo-Morales M. Telehealth system (e-CUIDATE) to improve quality of life in breast cancer survivors: rationale and study protocol for a randomized clinical trial. Trials. 2013 Jun 22;14:187. doi: 10.1186/1745-6215-14-187. PMID 23799886
- [Background] Ward EC, Sharma S, Burns C, Theodoros D, Russell T. Validity of conducting clinical dysphagia assessments for patients with normal to mild cognitive impairment via telerehabilitation. Dysphagia. 2012 Dec;27(4):460-72. doi: 10.1007/s00455-011-9390-9. Epub 2012 Jan 20. PMID 22271284
- [Background] Bedra M, McNabney M, Stiassny D, Nicholas J, Finkelstein J. Defining patient-centered characteristics of a telerehabilitation system for patients with COPD. Stud Health Technol Inform. 2013;190:24-6. PMID 23823363
- [Background] Bennell KL, Rini C, Keefe F, French S, Nelligan R, Kasza J, Forbes A, Dobson F, Abbott JH, Dalwood A, Vicenzino B, Harris A, Hinman RS. Effects of Adding an Internet-Based Pain Coping Skills Training Protocol to a Standardized Education and Exercise Program for People With Persistent Hip Pain (HOPE Trial): Randomized Controlled Trial Protocol. Phys Ther. 2015 Oct;95(10):1408-22. doi: 10.2522/ptj.20150119. Epub 2015 May 28. PMID 26023213
- [Background] Truter P, Russell T, Fary R. The validity of physical therapy assessment of low back pain via telerehabilitation in a clinical setting. Telemed J E Health. 2014 Feb;20(2):161-7. doi: 10.1089/tmj.2013.0088. Epub 2013 Nov 27. PMID 24283249
- [Background] Piqueras M, Marco E, Coll M, Escalada F, Ballester A, Cinca C, Belmonte R, Muniesa JM. Effectiveness of an interactive virtual telerehabilitation system in patients after total knee arthoplasty: a randomized controlled trial. J Rehabil Med. 2013 Apr;45(4):392-6. doi: 10.2340/16501977-1119. PMID 23474735
- [Background] Moffet H, Tousignant M, Nadeau S, Merette C, Boissy P, Corriveau H, Marquis F, Cabana F, Ranger P, Belzile EL, Dimentberg R. In-Home Telerehabilitation Compared with Face-to-Face Rehabilitation After Total Knee Arthroplasty: A Noninferiority Randomized Controlled Trial. J Bone Joint Surg Am. 2015 Jul 15;97(14):1129-41. doi: 10.2106/JBJS.N.01066. PMID 26178888
- [Background] Tousignant M, Giguere AM, Morin M, Pelletier J, Sheehy A, Cabana F. In-home telerehabilitation for proximal humerus fractures: a pilot study. Int J Telerehabil. 2015 Jan 29;6(2):31-7. doi: 10.5195/ijt.2014.6158. eCollection 2014 Fall. PMID 25945227
- [Background] Bedra M, Finkelstein J. Feasibility of post-acute hip fracture telerehabilitation in older adults. Stud Health Technol Inform. 2015;210:469-73. PMID 25991191
- [Background] Davidoff F, Batalden P, Stevens D, Ogrinc G, Mooney S; SQUIRE Development Group. Publication guidelines for quality improvement in health care: evolution of the SQUIRE project. Qual Saf Health Care. 2008 Oct;17 Suppl 1(Suppl_1):i3-9. doi: 10.1136/qshc.2008.029066. PMID 18836063
- [Background] 2011 ©WHO. International statistical classification of diseases and related health problems. - 10th revision, edition 2010. 3 v. Contents: v. 1. Tabular list - v. 2. Instruction manual - v. 3. Alphabetical index. 1.Diseases - classification. 2.Classification.
- [Background] Beaton DE, Richards RR. Measuring function of the shoulder. A cross-sectional comparison of five questionnaires. J Bone Joint Surg Am. 1996 Jun;78(6):882-90. doi: 10.2106/00004623-199606000-00011. PMID 8666606
- [Background] Dawson J, Doll H, Fitzpatrick R, Jenkinson C, Carr AJ. The routine use of patient reported outcome measures in healthcare settings. BMJ. 2010 Jan 18;340:c186. doi: 10.1136/bmj.c186. PMID 20083546
- [Background] Schmidt S, Ferrer M, Gonzalez M, Gonzalez N, Valderas JM, Alonso J, Escobar A, Vrotsou K; EMPRO Group. Evaluation of shoulder-specific patient-reported outcome measures: a systematic and standardized comparison of available evidence. J Shoulder Elbow Surg. 2014 Mar;23(3):434-44. doi: 10.1016/j.jse.2013.09.029. Epub 2014 Jan 7. PMID 24406123
- [Background] Muniz J, Elosua P, Hambleton RK; International Test Commission. [International Test Commission Guidelines for test translation and adaptation: second edition]. Psicothema. 2013;25(2):151-7. doi: 10.7334/psicothema2013.24. Spanish. PMID 23628527
- [Background] Membrilla-Mesa MD, Tejero-Fernandez V, Cuesta-Vargas AI, Arroyo-Morales M. Validation and reliability of a Spanish version of Simple Shoulder Test (SST-Sp). Qual Life Res. 2015 Feb;24(2):411-6. doi: 10.1007/s11136-014-0760-2. Epub 2014 Jul 20. PMID 25038636
- [Background] Angst F, Schwyzer HK, Aeschlimann A, Simmen BR, Goldhahn J. Measures of adult shoulder function: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) and its short version (QuickDASH), Shoulder Pain and Disability Index (SPADI), American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form, Constant (Murley) Score (CS), Simple Shoulder Test (SST), Oxford Shoulder Score (OSS), Shoulder Disability Questionnaire (SDQ), and Western Ontario Shoulder Instability Index (WOSI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S174-88. doi: 10.1002/acr.20630. No abstract available. PMID 22588743
- [Background] Roddey TS, Olson SL, Cook KF, Gartsman GM, Hanten W. Comparison of the University of California-Los Angeles Shoulder Scale and the Simple Shoulder Test with the shoulder pain and disability index: single-administration reliability and validity. Phys Ther. 2000 Aug;80(8):759-68. PMID 10911414
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738
- [Background] Roy JS, MacDermid JC, Woodhouse LJ. A systematic review of the psychometric properties of the Constant-Murley score. J Shoulder Elbow Surg. 2010 Jan;19(1):157-64. doi: 10.1016/j.jse.2009.04.008. PMID 19559630
- [Background] Castellet Feliu E 1, Vidal N 1 CX 2. Escalas de valoración en cirugía ortopédica y traumatología Rating scales in orthopaedic surgery and traumatology. Trauma Fund MAPFRE Vol 21 Supl 134-43.
- [Background] Conboy VB, Morris RW, Kiss J, Carr AJ. An evaluation of the Constant-Murley shoulder assessment. J Bone Joint Surg Br. 1996 Mar;78(2):229-32. PMID 8666631
- [Background] Livain T, Pichon H, Vermeulen J, Vaillant J, Saragaglia D, Poisson MF, Monnet S. [Intra- and interobserver reproducibility of the French version of the Constant-Murley shoulder assessment during rehabilitation after rotator cuff surgery]. Rev Chir Orthop Reparatrice Appar Mot. 2007 Apr;93(2):142-9. doi: 10.1016/s0035-1040(07)90217-2. French. PMID 17401287
- [Background] Bakken S, Grullon-Figueroa L, Izquierdo R, Lee NJ, Morin P, Palmas W, Teresi J, Weinstock RS, Shea S, Starren J; IDEATel Consortium. Development, validation, and use of English and Spanish versions of the telemedicine satisfaction and usefulness questionnaire. J Am Med Inform Assoc. 2006 Nov-Dec;13(6):660-7. doi: 10.1197/jamia.M2146. Epub 2006 Aug 23. PMID 16929036
- [Background] Demiris G, Speedie S, Finkelstein S. A questionnaire for the assessment of patients' impressions of the risks and benefits of home telecare. J Telemed Telecare. 2000;6(5):278-84. doi: 10.1258/1357633001935914. PMID 11070589
- [Background] Glick HA, Doshi JA, Sonnad SS PD. Economic Evaluation in Clinical Trials. 2nd edition. Oxford, UK: Oxford University Press; 2014.
- [Background] Tousignant M, Moffet H, Nadeau S, Merette C, Boissy P, Corriveau H, Marquis F, Cabana F, Ranger P, Belzile EL, Dimentberg R. Cost analysis of in-home telerehabilitation for post-knee arthroplasty. J Med Internet Res. 2015 Mar 31;17(3):e83. doi: 10.2196/jmir.3844. PMID 25840501
- [Background] Piaggio G, Elbourne DR, Altman DG, Pocock SJ, Evans SJ; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: an extension of the CONSORT statement. JAMA. 2006 Mar 8;295(10):1152-60. doi: 10.1001/jama.295.10.1152. PMID 16522836
- [Background] Bini SA, Mahajan J. Clinical outcomes of remote asynchronous telerehabilitation are equivalent to traditional therapy following total knee arthroplasty: A randomized control study. J Telemed Telecare. 2017 Feb;23(2):239-247. doi: 10.1177/1357633X16634518. Epub 2016 Jul 9. PMID 26940798
- [Background] Agostini M, Moja L, Banzi R, Pistotti V, Tonin P, Venneri A, Turolla A. Telerehabilitation and recovery of motor function: a systematic review and meta-analysis. J Telemed Telecare. 2015 Jun;21(4):202-13. doi: 10.1177/1357633X15572201. Epub 2015 Feb 22. PMID 25712109
- [Background] Tousignant M, Hamel M, Brière S. In-Home Telerehabilitation as an alternative to face-to-face treatment : Feasability in post-knee arthroplasty , speech therapy and Chronic Obstructive Pulmonary Disease.
- [Derived] Pastora-Bernal JM, Martin-Valero R, Baron-Lopez FJ, Garcia-Gomez O. Effectiveness of telerehabilitation programme following surgery in shoulder impingement syndrome (SIS): study protocol for a randomized controlled non-inferiority trial. Trials. 2017 Feb 23;18(1):82. doi: 10.1186/s13063-017-1822-x. PMID 28231815